CLINICAL TRIAL: NCT03169283
Title: Investigation of How Morning Nutrition Influences Cognitive Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PEP-1323
Record Dates: First submitted 2014-11-05; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Cognitive Performance
MeSH Terms: interventions — Edible Grain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cereal 1 (Experimental): A cereal high in viscous dietary fiber B glucan
  Interventions: Other: Cereal with B glucan
- Cereal 2 (Active Comparator): A cereal without B glucan
  Interventions: Other: Cereal without B glucan

INTERVENTIONS:
Other: Cereal with B glucan — A cereal high in viscous dietary fiber B glucan
  Arms: Cereal 1
Other: Cereal without B glucan — Cereal without B glucan
  Arms: Cereal 2

SUMMARY:
This project will assess the effects of the macro-nutrient make-up of morning food intake on cognitive performance using visual analog scale (VAS) measures, behavioral tests, and advanced high-density electrophysiological techniques (256-channel recordings). Two Isocaloric cereal products will be tested and compared to determine if measures of cognitive performance as well as satiety will change after consumption.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and taking no regular medications other than birth control or hormone replacement therapy
* Willing to use an effective contraceptive during the study, if sexually active and capable of bearing children
* Willing and able to sign informed consent
* Normal or corrected-to-normal vision
* Normal or corrected-to-normal hearing
* No history of neurological or psychiatric illness, including major depressive disorder and attention deficit disorder
* No history of substance, nicotine or alcohol dependence
* BMI below 35

Exclusion Criteria:

* Women who are pregnant or nursing
* Gain or loss of > 4kg in the last 3 months.
* Currently taking supplements or medications for weight loss
* Currently taking medications for neurological or psychiatric illness
* Diabetes mellitus (fasting glucose >126 mg/dL) or history of diabetes
* Dietary restraint on the Three Factor Eating Questionnaire score greater than or equal to 14
* Allergy to any of the foods used for the test breakfasts (oats or milk)
* History of GI disorders or GI surgical procedures for weight loss
* History of eating disorders
* Daily consumption of more than 400 mg of caffeine

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
cognitive performance | 0-4 hours
  cognitive performance using psychometric scales

SECONDARY OUTCOMES:
subjective measures of hunger | 0-4 hours
  subjective measures of hunger using Visual Analog Scale

CONTACTS AND LOCATIONS:
Overall Officials: John Foxe, PhD, Principal Investigator — The Sheryl and Daniel R. Tishman Cognitive Neurophysiology Laboratory
Locations (1):
- The Sheryl and Daniel R. Tishman Cognitive Neurophysiology Laboratory, The Bronx, New York, United States

REFERENCES:
- [Derived] Wilson TJ, Gray MJ, Van Klinken JW, Kaczmarczyk M, Foxe JJ. Macronutrient composition of a morning meal and the maintenance of attention throughout the morning. Nutr Neurosci. 2018 Dec;21(10):729-743. doi: 10.1080/1028415X.2017.1347998. Epub 2017 Jul 17. PMID 28714768